CLINICAL TRIAL: NCT06783790
Title: An Exploratory Clinical Study of the Safety and Efficacy of Avapritinib Combined With Azacitidine and Venetoclax in the Treatment of Relapsed Acute Myeloid Leukemia After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Avapritinib Combined With Azacitidine and Venetoclax in the Treatment of Relapsed AML After Allo-HSCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024097
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: AML (Acute Myelogenous Leukemia)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — avapritinib; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Avapritinib combined with Azacitidine and Venetoclax
  Interventions: Drug: Avapritinib, azacitidine, Venetoclax

INTERVENTIONS:
Drug: Avapritinib, azacitidine, Venetoclax — A: Induction therapy period: After patients were screened and enrolled, they began to receive 1-2 cycles of induction therapy, and the specific administration regimen was as follows: Avapritinib 100mg po qd D1-D14, azacitidine 35mg/m2 ih D1-D5, Venetoclax 100mg po qd D1-D14. The 28-day cycle was followed by curative effect evaluation at the end of each cycle. Patients who achieved complete remission entered the consolidation treatment stage.
  B: Consolidation therapy period: Patients who achieved complete remission after 1-2 cycles of induction therapy continued to receive avapritinib 100mg/d po. monotherapy for consolidation therapy, with a cycle of 28 days and a total of 4 cycles

SUMMARY:
This is a single-center, prospective, single-arm, exploratory clinical study. To explore the efficacy and safety of avapritinib in patients with recurrent acute myeloid leukemia after allogeneic hematopoietic stem cell transplantation with C-KIT mutation RUNX1::RUNX1T1 or CBFB::MYH11.

DETAILED DESCRIPTION:
We enrolled 20 patients with recurrent acute myeloid leukemia after allogeneic hematopoietic stem cell transplantation of RUNX1::RUNX1T1 or CBFB::MYH11 with C-KIT mutation.

The study was divided into induction therapy period and consolidation therapy period, and the study design was as follows:

A: Induction therapy period: After patients were screened and enrolled, they began to receive 1-2 cycles of induction therapy, and the specific administration regimen was as follows: Avapritinib 100mg po qd D1-D14, azacitidine 35mg/m2 ih D1-D5, Venetoclax 100mg po qd D1-D14. The 28-day cycle was followed by curative effect evaluation at the end of each cycle. Patients who achieved complete remission entered the consolidation treatment stage.

B: Consolidation therapy period: Patients who achieved complete remission after 1-2 cycles of induction therapy continued to receive avapritinib 100mg/d po. monotherapy for consolidation therapy, with a cycle of 28 days and a total of 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects met the criteria for recurrence after allogeneic transplantation: re-emergence of leukemia cells or bone marrow original cells in peripheral blood >5% (except for other causes such as bone marrow recovery period) or extramedullary leukemia cell infiltration or molecular or cytogenetic recurrence.
2. Bone marrow molecular biology detected C-KIT D816 or C-KIT N822 mutations
3. Patients with CBFB::MYH11 gene or RUNX1::RUNX1T1 fusion gene detected.
4. Eastern Cancer Collaboration Group (ECOG) physical status score 0-2 points.
5. Liver, kidney and cardiopulmonary functions met the following requirements: Within 2 weeks before enrollment ① creatinine ≤1.5 upper limit of normal value; ② Left ventricular ejection fraction ≥50%; ③ Blood oxygen saturation >91%; ④ Total bilirubin ≤2×ULN; ALT and AST≤2.5 x ULN; Myocardial enzymes < 2 times the upper limit of normal (for the same age)
6. Volunteer to participate in clinical studies and sign informed consent, willing to follow and able to complete all trial procedures.

Exclusion Criteria:

1. Known allergy to KIT inhibitor drug analogues.
2. Patients who have received previous treatment with Midostaurin.
3. Patients who have previously been treated with mutation-specific C-KIT inhibitors and have developed disease progression during treatment.
4. FLT3-ITD mutation in patients with recurrent/refractory disease (except low gene ratio).
5. HIV infected persons, HBV, HCV active infected persons.
6. Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases and other diseases.
7. With uncontrolled active GVHD (NIH for GVHD diagnosis and classification standards, aGVHD classification refer to the improved Glucksberg standard).
8. Central nervous system leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
2-month ORR after induction therapy | 2 months after induction therapy
  2-month objective remission rate after induction therapy

SECONDARY OUTCOMES:
CR rate after induction therapy | 2 months after induction therapy
  CR rate after 2 months
MRD negative rate after induction therapy | 2 months after induction therapy
  MRD negative rate after 2 months
Response rate after Consolidation treatment | 6 months after Consolidation treatment
  Response rate after 6 months
Safety | 2 years
  Types of adverse events (AE), AE severity, Relevance to study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Erlie Jiang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No